CLINICAL TRIAL: NCT02529579
Title: Safety and Efficacy Evaluation of iAPA-DC/CTL Combined Gemcitabine Therapy on Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: ImmunoGene Biotechology Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Zhaoshen Li, director of department of gastroenterology, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cellular immunotherapy
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: adoptive Cellular Immunotherapy; patient safety; therapeutic effect
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Gemcitabine (Active Comparator): Standard Gemcitabine Therapy
  Interventions: Drug: Gemcitabine
- cellular immunotherapy & Gemcitabine (Experimental): iAPA-DC/CTL adoptive cellular immunotherapy combined Standard Gemcitabine Therapy
  Interventions: Other: iAPA-DC/CTL adoptive cellular immunotherapy; Drug: Gemcitabine

INTERVENTIONS:
Other: iAPA-DC/CTL adoptive cellular immunotherapy — twice DC cell infusion and CTL cell infusion for 6 times
  Arms: cellular immunotherapy & Gemcitabine
Drug: Gemcitabine — standard Gemcitabine therapy

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of iAPA-DC/CTL combined gemcitabine therapy on advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced Pancreatic cancer patients with histological pathology confirmation
2. Both gender, aged 18-70 year-old
3. Bone marrow functioned well
4. Renal function normal
5. Liver function normal
6. patients are voluntary, and willing to sign informed consent
7. expected lifetime was at least 3 months

Exclusion Criteria:

1. With acute inflammation
2. Accompanied with primary malignant tumor other than pancreas
3. with autoimmune disease
4. using corticosteroid or other suppress immune hormone treatment
5. had transplant operation of vital organs
6. active hepatitis
7. HIV positive
8. dysfunction in blood coagulation
9. serious diseases in circulatory and respiratory systems
10. pregnancy or breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
6-month SR | 6 months
  6 months survival rate

SECONDARY OUTCOMES:
PFS | 6 months
  progression-Free Survival
OS | 6 months
  Over survival
ORR | 2 months
  Objective Response Rate
QOL | 2 months
  Quality of Life

OTHER OUTCOMES:
immunological markers | 2 months
  CD3, CD4,CD8,CD16,CD56,CD45,Treg(CD4,CD25, CD127low), IL-1B,IL-2R, IL-10,TNF-a，
Serum tumor biomarker | 2 months
  CA19-9,CEA

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Ii, MD, Principal Investigator — Changhai Hosptial,Second Military medical University
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China